CLINICAL TRIAL: NCT06806007
Title: Incentive Spirometer Training and Oropharyngeal Motor Training for Pulmonary Dysfunction in Spastic Diplegic Children
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Alaa Ebrahim Ahmed Mohammed Elshamy, Bachelor's degree, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KFSIRB200-342
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Dysfunction; Spastic Diaplegia
Keywords: Pulmonary dysfunction

STUDY DESIGN:
Intervention Model Description: Intervention study model Parallel assignment The study will include 48 spastic diplegic children suffering from pulmonarydysfunction ( age 3-7 years old )
  Children meeting the inclusion criteria will be randomly assigned to three experimental groups :
  First experimental group: children in this group will receive the incentive spirometer training Second experimental group: children in this group will receive oropharyngeal motor training Third experimental group: children in this group will receive a combination program of the incentive spirometer training and oropharyngeal motor training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A : Will include 16 spastic diplegic Children suffer from pulmonary dysfunction from both gend (Experimental): Each child in the group A will receive the incentive spirometer training , attending three sessions per week for three consecutive months. The duration of the session will be half an hour Set up
  1. Begin bothering child sit on the mat or chair.
  2. Hold the incentive spirometer in an upright position.
  3. The child Breathe out normally.
  4. Place the spirometer mouthpiece in child's mouth and ask him to close his / her lips tightly around it.
  5. Ask the child to Breathe in through mouth as slowly and deeply as he can,
  6. Hold breath for as long as possible, or at least five seconds. Exhale slowly
  7. Rest for a few seconds, and then repeat the first five steps at least 10 times every hour you're awake.
  8. After each set of 10 deep breaths, ask child cough deeply to clear lungs
  Interventions: Device: Group A
- Group B :Will include 16 spastic diplegic Children suffer from pulmonary dysfunction from both gende (Experimental): Each child in the group B will receive the oropharyngeal motor training programme , attending three sessions per week for three consecutive months. The duration of the session will be an hour The training programme consists of 10 individual mobilization exercises involving orofacial and pharyngeal area that required 45 minutes Each exercise had to be repeated for 10 times.
  The 10 exercises are:
  * Exercise 1: Pushing Up The Tongue
  * Exercise 2: Touching Nose
  * Exercise 3: Touching Chin
  * Exercise 4: Pushing Tongue Right and Left
  * Exercise 5: Folding Tongue
  * Exercise 6: Clicking the Tongue
  * Exercise 7: Pushing Tongue Against Spoon
  * Exercise 8: Holding A Spoon
  * Exercise 9: Holding Button with Lips
  * Exercise 10: Gargling
  Interventions: Other: Group B
- Group C : Will include 16 spastic diplegic Children suffer from pulmonary dysfunction from both gend (Experimental): Each child in the group C will receive a combination program of the incentive spirometer training and oropharyngeal motor training programme attending three sessions per week for three consecutive months. The duration of the session will be one hour and half that Will be designed into half an hour for the incentive spirometer training and an hour for the oropharyngeal motor training programme
  Interventions: Combination Product: Group C

INTERVENTIONS:
Device: Group A — Each child in the group A will receive the incentive spirometer training , attending three sessions per week for three consecutive months. The duration of the session will be half an hour Set up
  1. Begin bothering child sit on the mat or chair.
  2. Hold the incentive spirometer in an upright position.
  3. The child Breathe out normally.
  4. Place the spirometer mouthpiece in child's mouth and ask him to close his / her lips tightly around it.
  5. Ask the child to Breathe in through mouth as slowly and deeply as he can,
  6. Hold breath for as long as possible, or at least five seconds. Exhale slowly
  7. Rest for a few seconds, and then repeat the first five steps at least 10 times every hour you're awake.
  8. After each set of 10 deep breaths, ask child cough deeply to clear lungs
  Arms: Group A : Will include 16 spastic diplegic Children suffer from pulmonary dysfunction from both gend
Other: Group B — Each child in the group B will receive the oropharyngeal motor training programme , attending three sessions per week for three consecutive months. The duration of the session will be an hour The training programme consisted of 10 individual mobilization exercises involving orofacial and pharyngeal area that required 45 minutes Each exercise had to be repeated for 10 times.
  The 10 exercises are:
  * Exercise 1: Pushing Up The Tongue
  * Exercise 2: Touching Nose
  * Exercise 3: Touching Chin
  * Exercise 4: Pushing Tongue Right and Left
  * Exercise 5: Folding Tongue
  * Exercise 6: Clicking the Tongue
  * Exercise 7: Pushing Tongue Against Spoon
  * Exercise 8: Holding A Spoon
  * Exercise 9: Holding Button with Lips
  * Exercise 10: Gargling
  Arms: Group B :Will include 16 spastic diplegic Children suffer from pulmonary dysfunction from both gende
Combination Product: Group C — Each child in the group C will receive a combination program of the incentive spirometer training and oropharyngeal motor training programme attending three sessions per week for three consecutive months. The duration of the session will be one hour and half that Will be designed into half an hour for the incentive spirometer training and an hour for the oropharyngeal motor training programme
  Arms: Group C : Will include 16 spastic diplegic Children suffer from pulmonary dysfunction from both gend

SUMMARY:
Purpose of the study to determine the impact of incentive spirometer training and the oropharyngeal motor training or the combination of both for pulmonary dysfunction in spastic diplegic children

DETAILED DESCRIPTION:
This is a prospective randomized controlled clinical trial, conducted at Kafr El sheikh Hospital.

* Forty-eight children of both genders.
* The study will include children (age 3-7 years) post selective pulmonary dysfunction.
* Children meeting the inclusion criteria will be randomly assigned to one of three groups:
* first Experimental Group: children in this group will receive incentive spirometer training.
* second Experimental Group:children in this group will receive oropharyngeal motor training. .
* third experimental Group: Patients in this group will receive combination of incentive spirometer training and oropharyngeal motor training
* Randomization will be achieved using computer-generated random numbers to ensure an equal distribution of patients between the two groups.

Conditions: Cerebral Palsy

ELIGIBILITY:
Inclusion Criteria:

* the children with spastic CP between the age from 3 to 7 years old.

Level I to IV on the gross motor function classification system (GMFCS) , who have the partial ability to maintain antigravity head and trunk postures.

* Cognitive and cooperative function allowing pulmonary function measurements.
* No history of psychiatric or neurological disorders rather than cp.

Exclusion Criteria:

* Any uncontrolled clinically significant medical conditions such as coexistent cardiac disease or respiratory disease
* Children with cognitive impairment who are unable to comply with the protocol required procedure
* Children who are taking medications that can affect respiratory function
* Children with presence or history of tracheostomy

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
forced vital capacity (FVC) | Two months
  1) By using digital incentive spirometry which is the amount of air that an individual is able to forcibly exhale from his / her lungs after taking the deepest breath they can.
forced expiratory volume at 1 s (FEV1) | Two months
  1) By using digital incentive spirometry refers to the air an individual can exhale during a forced breath in 1 second
FVC/FEV1 ratio | Two months
  1) By using digital incentive spirometry refers to the air an individual can exhale during a forced breath in 1 second
expiratory reserve volume (ERV) | Two months
  1) By using digital incentive spirometry the amount of extra air above normal that you exhale during a forceful breath out.
Peak expiratory flow (PEF) | Two months
  the volume of air forcefully expelled from the lungs in one quick exhalation
forced expiratory flow (FEF) | Two months
  the speed that someone can breathe out air from their lungs, measured in the middle of a hard, fast breath out.
tidal volume (TV) | Two months
  refers to the air an individual can exhale during a forced breath in 1 second
inspiratory reserve volume (IRV) | Two months
  the additional volume of air that can be inspired at the end of a normal or tidal inspiration
the orofacial myofunctional clinical evaluation | Two months
  the OMES protocol is an instrument for the clinical evaluation of orofacial structures and functions of children that will permit the examiner to express numerically his perception of the characteristics and behaviors observed, and that can be administered without special equipment and in a brief manner

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of physical therapy Kafrelsheikh University, Kafrelsheikh, KafrelsheikhU
  - Faculty of physical therapy Kafrelsheikh University, Kafrelsheikh, Kafrelsheikh

IPD SHARING:
Plan to Share IPD: No